CLINICAL TRIAL: NCT00546273
Title: Double-Blind, Randomized, Placebo-Controlled Phase I Study, to Study the Tolerability and Immunogenicity of 4 RUTI Antituberculous Vaccine Different Doses (5, 25, 100 y 200µg of FCMtb) in Healthy Volunteers
Brief Title: Clinical Trial to Study 4 Different Doses of the Vaccine RUTI in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Archivel Farma S.L. (Industry)
Responsible Party: Pere-Joan Cardona, Fundacio Institut Germans Trias i Pujol
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FA/MI/01; EudraCT Number: 2006-000690-29
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Results first posted 2009-03-25 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Latent Tuberculosis Infection; Tuberculosis
Keywords: LTBI (Latent tuberculosis infection); TB(Tuberculosis); Vaccine
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- RUTI 5 micrograms of FCMtb (Experimental): RUTI dose: 5 micrograms of FCMtb (for fragmented cells of M. tuberculosis) (n=4)
  Interventions: Biological: RUTI
- RUTI 25 micrograms of FCMtb (Experimental): RUTI dose: 25 micrograms of FCMtb (for fragmented cells of M. tuberculosis) (n=4)
  Interventions: Biological: RUTI
- RUTI 100 micrograms of FCMtb (Experimental): RUTI dose: 100 micrograms of FCMtb (for fragmented cells of M. tuberculosis) (n=4)
  Interventions: Biological: RUTI
- RUTI 200 micrograms of FCMtb (Experimental): RUTI 200 micrograms of FCMtb (for fragmented cells of M. tuberculosis) (n=4)
  Interventions: Biological: RUTI
- placebo (Placebo Comparator): placebo of the vaccine RUTI (total n=8, n=2 for each period)
  Interventions: Biological: placebo of the vaccine RUTI

INTERVENTIONS:
Biological: RUTI — dose: 5 micrograms of FCMtb; given subcutaneously twice, on days 0 and 28
  Other Names: FCMtb is the active compound of the vaccine RUTI
  Arms: RUTI 5 micrograms of FCMtb
Biological: RUTI — dose: 25 micrograms of FCMtb; given subcutaneously twice, on days 0 and 28
  Other Names: FCMtb is the active compound of the vaccine RUTI
  Arms: RUTI 25 micrograms of FCMtb
Biological: RUTI — dose: 100 micrograms of FCMtb; given subcutaneously twice, on days 0 and 28
  Other Names: FCMtb is the active compound of the vaccine RUTI
  Arms: RUTI 100 micrograms of FCMtb
Biological: RUTI — dose: 200 micrograms of FCMtb; given subcutaneously twice, on days 0 and 28
  Other Names: FCMtb is the active compound of the vaccine RUTI
  Arms: RUTI 200 micrograms of FCMtb
Biological: placebo of the vaccine RUTI — placebo of the vaccine RUTI given subcutaneously twice, on days 0 and 28
  Other Names: placebo
  Arms: placebo

SUMMARY:
The aim of this study is to evaluate the safety of a new vaccine against Tuberculosis (RUTI) when administered to healthy adult volunteers, compared to placebo; and determine its safe dosage range. An initial evaluation of immune responses to the vaccine compared to placebo will also be undertaken.

In the present Phase I clinical trial, four increasing doses of RUTI will be tested, the groups composed by 6 volunteers each. (Total of 24 volunteers). The escalation to a new dose to test will be done after the safety of the previous dose has been ensured.

For each dose of FCMtb to test, each volunteer will be inoculated twice (at day 0 and day 28) with RUTI (4 volunteers) or placebo (2 volunteers) and will be followed-up up to 25 weeks from the first inoculation. The global length of the study will be approximately 15 months.

DETAILED DESCRIPTION:
RUTI is a therapeutic vaccine made from virulent M.tuberculosis bacteria, grown in stressful conditions, fragmented, detoxified, heat inactivated (FCMtb) and liposomed. RUTI provides a strong humoral and cellular immune response against antigens from active growing and latent bacilli but also against structural antigens, as it has been proved in animal models of latent tuberculosis infection. The vaccine has been designed to be used against Latent Tuberculosis Infection as a therapeutic vaccine after 1-month of chemotheraputic treatment, instead the current treatment based on 6-9 months of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy, based on medical examination at inclusion
* Male Caucasian subjects, aged between 18 and 40 years
* Willing and likely to be able to comply with the trial procedures

Exclusion Criteria:

* Evidence of previous, current or latent tuberculosis, as radiological findings on chest X ray compatible with previous or current infection with tuberculosis
* Positive T-SPOT TB result
* BCG-vaccinated subjects
* History of severe organ-system diseases, including
* History of allergic disorders or known hypersensitivity to any drug or vaccine, or to any of the vaccine to be studied components
* Personal or familiar history of autoimmune diseases, or Positive Antinuclear Antibodies
* HIV, HBV and HCV sero-positive
* Suspected or known current drug and/or alcohol abuse (as defined by an alcohol intake of > 50 g a day
* Lost of more than 400 mL of blood within 12 weeks, or more than 250 mL within 4 weeks, before the recruitment
* Laboratory parameters outside of normal ranges considered clinically significant
* Intake of trial medication in other clinical trials within 1 month of the first vaccination
* Intake of any other drugs that could not be eliminated of the body before the first vaccination, especially anti-inflammatory nonsteroid and corticosteroid drugs
* Acute disease with > 37ºC temperature within 72 hours before the first vaccination

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pere-Joan Cardona, MD, PhD, Principal Investigator — Unitat de Tuberculosi Experimental. Fundació Institut per la Investigació en Ciències de la Salut Germans Trias i Pujol.; Joan Costa, MD, PhD, Principal Investigator — Pharmacology Department. Hospital Universitari "Germans Trias i Pujol"
Locations (3):
- Spain (3):
  - Experimental Tuberculosis Unit. Fundació Institut per la Investigació Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Pharmacology Department. Hospital Universitari Germans Trias i Pujol., Badalona, Barcelona

REFERENCES:
- [Background] Cardona PJ, Amat I, Gordillo S, Arcos V, Guirado E, Diaz J, Vilaplana C, Tapia G, Ausina V. Immunotherapy with fragmented Mycobacterium tuberculosis cells increases the effectiveness of chemotherapy against a chronical infection in a murine model of tuberculosis. Vaccine. 2005 Feb 3;23(11):1393-8. doi: 10.1016/j.vaccine.2004.09.008. PMID 15661388
- [Background] Cardona PJ, Amat I. [Origin and development of RUTI, a new therapeutic vaccine against Mycobacterium tuberculosis infection]. Arch Bronconeumol. 2006 Jan;42(1):25-32. doi: 10.1016/s1579-2129(06)60110-9. Spanish. PMID 16426520
- [Background] Cardona PJ. RUTI: a new chance to shorten the treatment of latent tuberculosis infection. Tuberculosis (Edinb). 2006 May-Jul;86(3-4):273-89. doi: 10.1016/j.tube.2006.01.024. Epub 2006 Mar 20. PMID 16545981
- [Background] Vilaplana C, Ruiz-Manzano J, Gil O, Cuchillo F, Montane E, Singh M, Spallek R, Ausina V, Cardona PJ. The tuberculin skin test increases the responses measured by T cell interferon-gamma release assays. Scand J Immunol. 2008 Jun;67(6):610-7. doi: 10.1111/j.1365-3083.2008.02103.x. Epub 2008 Apr 4. PMID 18397200
- [Background] Guirado E, Gil O, Caceres N, Singh M, Vilaplana C, Cardona PJ. Induction of a specific strong polyantigenic cellular immune response after short-term chemotherapy controls bacillary reactivation in murine and guinea pig experimental models of tuberculosis. Clin Vaccine Immunol. 2008 Aug;15(8):1229-37. doi: 10.1128/CVI.00094-08. Epub 2008 Jun 4. PMID 18524883
- [Background] Gil O, Vilaplana C, Guirado E, Diaz J, Caceres N, Singh M, Cardona PJ. Enhanced gamma interferon responses of mouse spleen cells following immunotherapy for tuberculosis relapse. Clin Vaccine Immunol. 2008 Nov;15(11):1742-4. doi: 10.1128/CVI.00255-08. Epub 2008 Sep 30. PMID 18827194
- See also: Fundació Institut d'Investigació en Ciències de la Salut Germans Trias i Pujol homepage — http://www.germanstrias.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four RUTI doses were tested, in a sequencial way (n=6 each). 14 days before starting each level of treatment, subjects, after signing the informed consent, were screened in the Phase 1 Unit (Hospital Germans Trias i Pujol) in order to decide if they were elegible to be part of the study.
Pre-assignment Details: 24 volunteers were enrolled and distributed in 4 groups, one group for every period (each period: 6 new volunteers). There was one period per dose tested, and doses were tested increasingly, not beginning to test one dose until clinically ensured the safety of the previous dose. The double blind was opened at the end of the study.
Groups:
- RUTI 5 Micrograms of FCMtb: RUTI dose: 5 micrograms of FCMtb
- RUTI 25 Micrograms of FCMtb: RUTI dose: 25 micrograms of FCMtb
- RUTI 100 Micrograms of FCMtb: RUTI dose: 100 micrograms of FCMtb
- RUTI 200 Micrograms of FCMtb: RUTI dose: 200 micrograms of FCMtb
- Placebo: placebo of the vaccine RUTI, given subcutaneously twice, on days 0 and 28
Period: I
Arm/Group | RUTI 5 Micrograms of FCMtb | RUTI 25 Micrograms of FCMtb | RUTI 100 Micrograms of FCMtb | RUTI 200 Micrograms of FCMtb | Placebo
Started | 4 | 0 | 0 | 0 | 2
Completed | 4 | 0 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0
Period: II
Arm/Group | RUTI 5 Micrograms of FCMtb | RUTI 25 Micrograms of FCMtb | RUTI 100 Micrograms of FCMtb | RUTI 200 Micrograms of FCMtb | Placebo
Started | 0 | 4 | 0 | 0 | 2
Completed | 0 | 4 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0
Period: III
Arm/Group | RUTI 5 Micrograms of FCMtb | RUTI 25 Micrograms of FCMtb | RUTI 100 Micrograms of FCMtb | RUTI 200 Micrograms of FCMtb | Placebo
Started | 0 | 0 | 4 | 0 | 2
Completed | 0 | 0 | 4 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0
Period: IV
Arm/Group | RUTI 5 Micrograms of FCMtb | RUTI 25 Micrograms of FCMtb | RUTI 100 Micrograms of FCMtb | RUTI 200 Micrograms of FCMtb | Placebo
Started | 0 | 0 | 0 | 4 | 2
Completed | 0 | 0 | 0 | 4 | 2
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RUTI 5 Micrograms of FCMtb | RUTI 25 Micrograms of FCMtb | RUTI 100 Micrograms of FCMtb | RUTI 200 Micrograms of FCMtb | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.25 (2.87) | 26 (2.94) | 23 (2.16) | 22.25 (2.22) | 24 (4.75) | 24.08 (3.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 4 | 4 | 4 | 8 | 24
Region of Enrollment [Number; unit: participants]
  Spain | 4 | 4 | 4 | 4 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: VAS Pain Score (Visual Analogic Scale, That Ranges From 0 to 100) to Evaluate Each Volunteer Subjective Pain Intensity at the Inoculation Point
Time Frame: at protocol defined timepoints: days 0, 1, 3, 7, 21, 28, 29, 31, 35, 56
Reporting Status: Not Posted, anticipated posting 2008-11
Measure: Mean (Standard Deviation); unit: units on a scale

2. Secondary Outcome: Evaluation of the Immunogenicity of the Different Doses of the Vaccine Tested
Description: Immunological assays are performed at all timepoints to determine vaccine immunogenicity
Time Frame: at protocol defined timepoints: days 0, 7, 21, 28, 35, 56, 112 & 156
Reporting Status: Not Posted, anticipated posting 2008-11
Measure: Number (Standard Deviation)

3. Primary Outcome: Occurrence, Intensity and Relationship to Vaccination of Local and Systemic Events
Time Frame: during the whole study
Reporting Status: Not Posted, anticipated posting 2008-11
Measure: Number; unit: ocurrences/subjects (O/S)

4. Primary Outcome: Number of Clinically Relevant Abnormalities in the Laboratory Tests According to the Doctors' Impression
Description: haematological and biochemical laboratory tests
Time Frame: at protocol defined timepoints: days 0, 7, 21, 28, 35, 56, 112 & 156
Population: All the participants of the study were analyzed for this specific outcome measure.
Measure: Number; unit: number of abnormalities
Arm/Group | RUTI 5 Micrograms of FCMtb | RUTI 25 Micrograms of FCMtb | RUTI 100 Micrograms of FCMtb | RUTI 200 Micrograms of FCMtb | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8
number of abnormalities | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure of the results has to be previously arranged if mutually agreeable to both investigators and the company manufacturer of the vaccine RUTI: Archivel Farma S.L.